CLINICAL TRIAL: NCT04810026
Title: Transform Type 2: Examining How Meal-Delivery and Education Resources Affect Prediabetes and Type 2 Diabetes Symptoms and Self-Care
Brief Title: Transform Type 2: Examining Meal-Delivery and Education for Diabetes Self-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UnitedHealth Group (Industry)
Responsible Party: Principal Investigator, Shane Hoversten, Senior Research Fellow, UnitedHealth Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0068
Record Dates: First submitted 2021-03-12; First posted 2021-03-22 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: PreDiabetes; Diabetes Mellitus, Type 2
Keywords: diabetes mellitus, type 2; information seeking behavior; waist-hip ratio; blood pressure; weight; prediabetes; glycemic control; diet; life style; cholesterol; meal delivery; nutrition; continuous glucose monitoring; CGM; self report; education; coaching; yoga; meditation; human
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Information Seeking Behavior; Body Weight | interventions — Educational Status; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Education only (Active Comparator): Push notifications for online diabetes self-management education for 12 weeks, passive access to lifestyle education for 16 weeks
  Interventions: Behavioral: Education
- Group 2: Education and Meals (Experimental): Meal delivery (3 meals per day, 5 days per week) for 12 weeks, push notifications for online diabetes self-management education for 12 weeks, passive access to lifestyle education for 16 weeks
  Interventions: Behavioral: Education; Behavioral: Meal delivery
- Group 3: Education, Meals, Coaching (Experimental): Meal delivery (3 meals per day, 5 days per week) for 12 weeks, coaching program (e.g., diabetes-specific coaching and education, push notifications for lifestyle education modules, community support) for 12 weeks, and passive access to lifestyle education for final 4 weeks
  Interventions: Behavioral: Education; Behavioral: Meal delivery; Behavioral: Lifestyle coaching

INTERVENTIONS:
Behavioral: Education — Healthy-lifestyle and diabetes-related virtual education (text and videos)
  Other Names: diabetes self-management education; healthy-lifestyle education
Behavioral: Meal delivery — breakfast, lunch, and dinner adhering to the longevity diet macro-nutrient profiles
  Other Names: Nutrition for Longevity meals; Longevity Diet
  Arms: Group 2: Education and Meals; Group 3: Education, Meals, Coaching
Behavioral: Lifestyle coaching — calls with coach and/or nutritionist, access to Facebook community support group
  Other Names: Longevity Program
  Arms: Group 3: Education, Meals, Coaching

SUMMARY:
The purpose of this research is to understand the impact of medically tailored meals on health-related biometrics (e.g., glucose time-in-range, waist-hip ratio, cholesterol) and how providing medically tailored meals promotes engagement in diabetes education and drives information-seeking behavior.

DETAILED DESCRIPTION:
The purpose of this research is to understand the impact of medically tailored meals on health-related biometrics (e.g., glucose time-in-range, waist-hip ratio) and how providing medically tailored meals promotes engagement in diabetes education and drives information-seeking behavior. Secondary purposes are to characterize the relationship between information-seeking behaviors and glycemic control; to characterize the relationship between psychometric survey results and program engagement, biometrics, and information-seeking behaviors; and to understand how meal provision and materials influence program satisfaction and adherence to healthy diabetes-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient, employee, or employee dependent at Utica Park Clinic in Oklahoma
* Be diagnosed with type 2 diabetes, prediabetes, and/or have an A1c result of 5.7 percent or above
* Be above an ideal weight (for example, body mass index [BMI] greater than or equal to 25)
* 18 years of age or older
* Have UnitedHealthcare insurance for 1 year+
* Have an active e-mail address
* Have a smartphone with access to the internet that is compatible with the Dexcom G6 app

Exclusion Criteria:

* Be undergoing any form of cancer treatment
* Be pregnant or breastfeeding
* Have allergies to nightshade vegetable (e.g., bell peppers, potatoes, tomatoes) or legumes (e.g., green beans, peas), or tree nuts
* Currently taking anti-psychotic medications to control schizophrenia and bipolar disorders, as well as other mental disorders including dementia, major depression, and even drug addiction
* Be currently taking insulin
* Be currently taking sulfonylureas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Change in mean glucose time in range from baseline at Week 6 | Week 0 and Week 6
  Percentage of time estimated glucose value (EGV) from continuous glucose monitor (CGM) is between 70 mg/dL and 180 mg/dL, measured daily with weekly composite results
Change in mean glucose time in range from baseline at Week 12 | Week 0 and Week 12
  Percentage of time estimated glucose value (EGV) from CGM is between 70 mg/dL and 180 mg/dL, measured daily with weekly composite results
Change in mean glucose time in range from baseline at Week 16 | Week 0 and Week 16
  Percentage of time estimated glucose value (EGV) from CGM is between 70 mg/dL and 180 mg/dL, measured daily with weekly composite results

SECONDARY OUTCOMES:
Change in CGM-derived glucose features from baseline | Week 0, Week 6, Week 12, and Week 16
  Average of EGVs, percentage time above and below range (< 70 mg/dL or >180 mg/dL), and glucose variability (standard deviation of EGVs), measured via daily with weekly composite results
Change in blood test results from baseline | Week 0, Week 12
  Difference in measurements of HbA1c, HDL cholesterol, total cholesterol, LDL cholesterol, triglycerides, and high-sensitivity C-reactive protein (hs-CRP) obtained from blood tests
Change in self-reported waist-to-hip ratio | Weekly, Weeks 0-12
  waist circumference, hip circumference, self-reported weekly; calculated by dividing the waist circumference by the hip circumference
Change in self-reported blood pressure | Weekly, Weeks 0-12
  blood pressure, self-reported weekly

OTHER OUTCOMES:
Visits to site | Week 16
  Usage stats from website that hosts educational materials, from Week 1 through Week 16
Percentage of tasks completed | Week 16
  Usage stats from website that hosts educational materials, from Week 1 through Week 16
Number of interactions with lifestyle coach | Week 12
  Count of total interactions from Week 1 to Week 12
Change from baseline in modified Yale Food Addiction Scale score at Week 6, Week 13 | Week 0, Week 6, Week 13
  modified food addiction scale, compared to responses at baseline, where higher scoring indicate a worse outcome; to meet the food addiction threshold, participants must meet the threshold for either question 6 or 7, and the threshold for 3 or more of the remaining questions
Change from baseline in abbreviated Medical Outcomes Study Sleep Scale | Week 0, Week 13
  Responses to an abbreviated Medical Outcomes Study Sleep Scale, compared to responses at baseline; with the exception of question 2, higher scores indicate a worse outcome and the range of scores (excluding question 2) is 11 - 65

CONTACTS AND LOCATIONS:
Overall Officials: Katlyn A Fleming, PhD, Principal Investigator — UnitedHealth Group
Locations (1):
- OptumLabs, Minnetonka, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data (IPD) that has been collected during the trial and de-identified
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication, no end date
Access Criteria: Investigators who provide a methodologically sound proposal for analyses within the bounds of consent, and approved by an independent review committee for analyses not within the bounds of consent. Data will be stored in UnitedHealth Group database and will not be publicly available.